CLINICAL TRIAL: NCT05172505
Title: Transcranial Direct Current Stimulation in a Home Treatment Setting for Major Depression: A Double-blind, Placebo-controlled Pilot Trial
Brief Title: Transcranial Direct Current Stimulation in a Home Treatment Setting for Major Depression
Acronym: HomeDC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Daniel Keeser, Research Group Leader Neuromodulation And Multimodal NeuroImaging, Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HomeDC
Record Dates: First submitted 2021-10-20; First posted 2021-12-29 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Depression
Keywords: tDCS; Depression; Home Treatment
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active prefrontal tDCS 2mA 6 weeks 5x/week (Active Comparator)
  Interventions: Device: prefrontal tDCS
- Sham prefrontal tDCS 6 weeks 5x/week (Sham Comparator)
  Interventions: Device: prefrontal tDCS

INTERVENTIONS:
Device: prefrontal tDCS — 2 mA prefrontal tDCS (anode over F3, cathode over F4 10/20 EEG System) for 6 weeks, 5x/week in a home treatment Setting (self application) for 30 mins.

SUMMARY:
Non-invasive transcranial brain stimulation (NTBS) techniques are well established in experimental neuroscience and have been increasingly used in the treatment of mental illnesses, especially depressive disorders, in the last years. Transcranial direct current stimulation (tDCS) of prefrontal cortex regions has been reported to exert antidepressant effects. Treatment with tDCS for MDD requires sessions several times a week, which is very time-consuming and stressful for patients, as they have to come to the clinic almost every day. At the same time, the availability of non-drug therapies for MDD is limited, especially in more rural areas. The home-treatment approach with tDCS for MDD could address this problem and is of increasing interest in times of the Covid-19 pandemic, when frequent clinic visits should be avoided.

There are some studies on the home-treatment approach with tDCS for different, mainly neurological disorders such as parkinson's disease, multiple sclerosis and chronic pain. For the treatment of MDD with tDCS in the home treatment setting, only one pilot study has been published so far, which shows good feasibility and good antidepressant effects. However, this study does not include a placebo condition.

The study will be conducted in a double-blind, placebo-controlled, parallel-group design with 16 patients per group. Patients with MDD do a 6-weeks self-administered treatment with prefrontal tDCS (anode: F3, cathode: F4, 5 sessions/week, 30min/day, 2mA intensity) or sham tDCS (parameters correspondent active tDCS, ramp in and ramp out periods only without intermittent stimulation) as adjunctive treatment to a serotonergic medication or alone. For the continuous monitoring of the technical parameters and thus for quality control and for blinding, the same technical achievements as in the DepressionDC trial are used. As a new feature, a cap is used for easier handling in the home-treatment setting, in which electrodes are already integrated at the F3 and F4 points.

This study aims to investigate the feasibility and effectiveness of 6 weeks of daily home treatment with tDCS for MDD. According to the DepressionDC trial, the primary outcome parameters are the decrease in the MADRS after 6 weeks and at the end of the follow-up phase, as well as the feasibility based on the dropout rates and the outcome in the comfort rating questionnaire. Additional baseline examinations with cMRI and e-field modelling will investigate the possible influence of the individual e-field on the outcome.

DETAILED DESCRIPTION:
Design:

The study will be conducted in a double-blind, placebo-controlled, parallel-group design with 16 patients per group. Patients with primary diagnosis of MDD according to DSM-5 perform a 6-weeks self-administered treatment with prefrontal tDCS (anode over F3, cathode over F4, 5 sessions/week, 30min/day, 2mA intensity) or sham-tDCS (parameters correspondent active tDCS, ramp-in and ramp-out periods only without intermittent stimulation) as adjunctive treatment to a stable antidepressant medication or alone. The study will be conducted at the Department of Psychiatry and Psychotherapy of the LMU Munich. Suitable patients will be randomized into two groups after they passed screening. Stratification according to the severity of the depressive symptoms (MARDS<21 vs. MARDS≥21) to distribute patients according to factors influencing the clinical outcome will be also done as well as stratification according to gender. The groups will receive active tDCS or sham-tDCS for a total of 6 weeks (5x/week, 30 min. stimulation). At baseline, an optional baseline cMRI examination with e-field modelling and fMRI will be performed. During the treatment phases, a study visit will take place every 2 weeks. In addition, a study visit will take place after the first week to address any difficulties with self-application at home. After 6 weeks, the primary endpoint will be reached and a final rating will be made after the treatment phase. In the subsequent follow-up phase, a study visit (V5 and V6) will take place 4 weeks and 8 weeks after the last stimulation session. According to the rules of the DepressionDC trial (Padberg et al., 2017) a total of 4 sessions may be missed without a drop out. Missed sessions can be compensated with additional sessions in week 7. This yields a total of 6 study visits with a total protocol duration of 14 weeks. The treatment phase is 6 weeks long with a maximum of 30 tDCS sessions per patient in home treatment.

Patients which continue to have relevant depressive symptoms after the 6 weeks of active or sham tDCS and after completion of the follow up phase will be offered 6 weeks of active treatment after V5. Patients receiving the active phase after V5 will receive an additional 3 study visits with the same scales reported like V1/V2/V3 during this second study phase: V6 after the first 3 weeks of active treatment, V7 after 6 weeks and V8 as a follow up 4 weeks after completion of the second treatment phase. Effects of this second study phase will be analysed in an exploratory way on an intraindividual level.

ELIGIBILITY:
Inclusion Criteria:

* Primary DSM-5 diagnosis of Major Depression as assessed by the M.I.N.I with a single or recurrent episode with the additional requirements of a current episode with a duration of ≥4 weeks.
* Current depressive episode is less than 5 years duration (the definition of an episode is demarcated by a period of ≥2 months in which the patient did not meet full criteria for the DSM-5 definition of major depressive episode).
* Total HDRS-21 ≥13 at the screening visit.
* Patient is taking one of the following antidepressants of adequate dose and ≥2 weeks in the current Episode: SSRIs: Escitalopram, Citalopram, Sertralin, Paroxetin, Fluoxetin, Fluvoxamin; SSNRIs: Duloxetin, Venlafaxin, Milnacipran. and optional concomitant treatment with Quetiapin, Lithium und Mirtazapin.
* Capable and willing to provide informed consent.
* Negative pregnancy test and willingness to use contraceptive measures during study treatment for women with childbearing potential (i.e <. 2 years post-menopausal)

Exclusion Criteria:

* Investigators, site personnel directly affiliated with this study, and their immediate families
* Acute risk for suicide (MADRS, item 10 score of ≥4 or suicidal attempt in the present episode
* Treatment with electroconvulsive therapy in the present episode.
* Treatment with deep brain stimulation or vagus nerve stimulation and/or any other intracranial implants (clips, cochlear implants).
* Any other relevant psychiatric axis-I- and/or axis-II-disorder.
* Any relevant instable medical condition.
* Individuals diagnosed with a significant neurological disorder or insult including, but not limited to:

  * Increased intracranial pressure
  * Space occupying brain lesion
  * History of cerebrovascular accident
  * Transient ischemic attack within two years
  * Cerebral aneurysm, dementia
  * Parkinson's disease
  * Huntington's chorea
  * Multiple sclerosis
  * Epilepsy
* History of seizures
* Pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility | 6 weeks
  Drop out rates, number of completed stimulation sessions in the treatment phase

SECONDARY OUTCOMES:
Safety | 6 weeks
  side effects and complications encountered, rates of discontinuation of stimulations due to high impedances, number of SAEs and AEs
Change in BDI, GAF and CGI | 10 weeks
  The change in absolute score in the BDI, CGI and GAF after 6 weeks of tDCS treatment and after 4 weeks of follow up compared to the baseline scores
Change from baseline in the Montgomery Åsberg Depression Rating Scale (MADRS) scores at week 6 post-randomization compared to baseline | 6 weeks
  The change in absolute score in the MADRS after 6 weeks of tDCS treatment compared to the baseline MADRS score

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry and Psychotherapy, Ludwig-Maximilian University Munich, Munich, Germany

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Kumpf U, Ezim H, Stadler M, Burkhardt G, Palm U, Dechantsreiter E, Padberg F. Transcranial direct current stimulation as treatment for major depression in a home treatment setting (HomeDC trial): study protocol and methodology of a double-blind, placebo-controlled pilot study. Pilot Feasibility Stud. 2023 Dec 15;9(1):197. doi: 10.1186/s40814-023-01423-x. PMID 38102647
- [Derived] Kumpf U, Palm U, Eder J, Ezim H, Stadler M, Burkhardt G, Dechantsreiter E, Padberg F. TDCS at home for depressive disorders: an updated systematic review and lessons learned from a prematurely terminated randomized controlled pilot study. Eur Arch Psychiatry Clin Neurosci. 2023 Oct;273(7):1403-1420. doi: 10.1007/s00406-023-01620-y. Epub 2023 May 16. PMID 37191697